CLINICAL TRIAL: NCT04493853
Title: A Phase III Double-Blind, Randomised, Placebo-Controlled Study Assessing the Efficacy and Safety of Capivasertib+Abiraterone Versus Placebo+Abiraterone as Treatment for Patients With DeNovo Metastatic Hormone-Sensitive Prostate Cancer Characterised by PTEN Deficiency.
Brief Title: Capivasertib+Abiraterone as Treatment for Patients With Metastatic Hormone-sensitive Prostate Cancer and PTEN Deficiency
Acronym: CAPItello-281
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D361BC00001; 2023-504998-20-00 (Registry Identifier: CTIS); 2020-000346-33 (EudraCT Number)
Record Dates: First submitted 2020-07-09; First posted 2020-07-30 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Hormone-Sensitive Prostate Cancer
Keywords: Prostate cancer; De Novo Metastatic Prostate cancer; PTEN; PTEN deficiency; Hormones; Hormone-Sensitive; Androgen Deprivation Therapy; Capivasertib; Abiraterone
MeSH Terms: conditions — Prostatic Neoplasms | interventions — capivasertib; Abiraterone Acetate

STUDY DESIGN:
Intervention Model Description: Approximately 1000 participants are assigned to one of the two parallel groups (1:1 ratio) to receive either capivasertib or placebo, in combination with abiraterone on a background of ADT for the duration of the study.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Capivasertib + Abiraterone (Experimental): Participants receive capivasertib in combination with abiraterone (prednisone/prednisolone) on a background of ADT.
  Interventions: Drug: Capivasertib; Drug: Abiraterone Acetate
- Placebo + Abiraterone (Placebo Comparator): Participants receive placebo in combination with abiraterone (prednisone/prednisolone) on a background of ADT.
  Interventions: Other: Placebo; Drug: Abiraterone Acetate

INTERVENTIONS:
Drug: Capivasertib — 400 mg (2 tablets) BD given on an intermittent weekly dosing schedule. Patients will be dosed on Days 1 to 4 in each week of a 28-day treatment cycle. Number of Cycles: until disease progression or unacceptable toxicity develops.
  Arms: Capivasertib + Abiraterone
Other: Placebo — matched to capivasertib appearance (2 tablets) BD given on an intermittent weekly dosing schedule. Patients will be dosed on Days 1 to 4 in each week of a 28-day treatment cycle. Number of Cycles: until disease progression or unacceptable toxicity develops.
  Arms: Placebo + Abiraterone
Drug: Abiraterone Acetate — Administered orally as tablets at a dosage of 1000 mg daily. Administered continuously until criteria for discontinuation are met.
  Other Names: ZYTIGA; Novadoz

SUMMARY:
This study will assess the efficacy and safety of capivasertib plus abiraterone (+prednisone/prednisolone) plus androgen deprivation therapy (ADT) versus placebo plus abiraterone (+prednisone/prednisolone) plus ADT in participants with mHSPC whose tumours are characterised by PTEN deficiency. The intention of the study is to demonstrate that in participants with mHSPC, the combination of capivasertib plus abiraterone (+prednisone/prednisolone) plus ADT is superior to placebo plus abiraterone (+prednisone/prednisolone) plus ADT in participants with mHSPC characterised by PTEN deficiency with respect to radiographic progression-free survival (rPFS) per 1) Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 for soft tissue and/or Prostate Cancer Working Group (PCWG3) for bone as assessed by the investigator 2) death due to any cause.

ELIGIBILITY:
Inclusion Criteria:

* Asymptomatic or mildly symptomatic, histologically-confirmed de novo hormone-sensitive prostate adenocarcinoma without small-cell tumours diagnosed within 180 days of randomisation
* Consent to provide a FFPE tissue block (preferred) or slides. Tissue from bone metastases is not acceptable
* A valid PTEN IHC result indicating PTEN deficiency (centralized testing)
* Metastatic disease documented prior to randomisation by clear evidence of ≥ 1 bone lesion and/or ≥ 1 soft tissue lesion accurately assessed at baseline and suitable for repeated assessment with CT and/or MRI. PSMA PET identification only will not be eligible
* Candidate for abiraterone and steroid therapy
* Ongoing ADT with GnRH analogue, or LHRH agonists or antagonist, or bilateral orchiectomy (regardless of method) is from 0 days to a max. of 93 days prior to randomisation
* Eastern Cooperative Oncology Group (ECOG)/WHO performance status 0 to 1 with no deterioration over the previous 2 weeks and minimum life expectancy of 12 weeks
* Able and willing to swallow and retain oral medication
* 7-day Brief Pain Inventory-Short Form (BPI-SF) and Brief Fatigue Inventory(BFI) questionnaires and the analgesic diary during screening completed. Participants must complete a minimum of 4 successful assessments within a 7-day period prior to randomisation.
* Agreement to remain abstinent (refrain from heterosexual intercourse) or use contraceptive measures, and agreement to refrain from donating sperm
* Capable of giving signed informed consent
* Provision of signed and dated written Optional Genetic Research Information informed consent prior to collection of samples

Exclusion Criteria:

* Prior radical prostatectomy or definitive radiotherapy with therapeutic intent for prostate cancer. Palliative radiotherapy is allowed providing any wide field radiation therapy is completed more than 4 weeks before the start of study treatment
* Major surgery (excluding placement of vascular access, transurethral resection of prostate, bilateral orchiectomy, or internal stents) within 4 weeks of the start of study treatment
* Brain metastases, or spinal cord compression (unless spinal cord compression is asymptomatic, treated and stable and not requiring steroids for at least 4 weeks prior to start of study treatment)
* Past medical history of interstitial lung disease, drug-induced interstitial lung disease, radiation pneumonitis which required steroid treatment, or any evidence of clinically active interstitial lung disease
* Any of the following cardiac criteria:

  i. Mean resting corrected QT interval (QTc) > 470 msec obtained from triplicate ECGs ii. History of QT prolongation associated with other medications that required discontinuation of that medication.

iii. Family history of long QT syndrome, or unexplained sudden death under 40 years of age in first-degree relatives.

iv. Medical history significant for arrhythmia which is symptomatic or requires treatment, symptomatic or uncontrolled atrial fibrillation despite treatment, or asymptomatic sustained ventricular tachycardia.

v. Any clinically important abnormalities in conduction or morphology of resting ECG (eg, complete left bundle branch block, third-degree heart block) vi. Any factors that increase the risk of QTc prolongation or risk of arrhythmic events such as hypokalaemia, potential for torsades de pointes, congenital long QT syndrome, or any concomitant medication known to significantly prolong the QT interval vii. Experience of any of the following procedures or conditions in the preceding 3 months: coronary artery bypass graft, angioplasty, myocardial infarction, angina pectoris.

viii. Congestive heart failure NYHA Grade ≥ 2 ix. Symptomatic hypotension - systolic blood pressure (SBP) <90 mmHg and/or diastolic blood pressure (DBP) <50 mmHg x. Uncontrolled hypertension (SBP ≥ 160 mmHg or DBP ≥ 95 mmHg).

* Clinically significant abnormalities of glucose metabolism as defined by any of the following:

  i. Patients with diabetes mellitus type 1 or diabetes mellitus type 2 requiring insulin treatment ii. HbA1c ≥8.0% (63.9 mmol/mol)
* Inadequate bone marrow reserve or organ function as demonstrated by any of the following laboratory values:

  i. Absolute neutrophil count < 1.5x 10^9/L ii. Platelet count < 100x 10^9/L iii. Haemoglobin < 9 g/dL (< 5.59 mmol/L) iv. Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) > 2.5x upper limit of normal (ULN) if no demonstrable liver metastases or > 5x ULN in the presence of liver metastases. Elevated alkaline phosphatase (ALP) is not exclusionary if due to the presence of bone metastases and liver function is otherwise considered adequate in the investigator's judgement v. Total bilirubin > 1.5x ULN (participants with confirmed Gilbert's syndrome may be included in the study with a higher value) vi. Creatinine clearance < 50 mL/min (measured or calculated by Cockcroft and Gault equation)
* As judged by the investigator, any evidence of severe or uncontrolled systemic diseases, including active bleeding diatheses, or known active infection including hepatitis B, hepatitis C, and HIV
* unevaluable for both bone and soft tissue progression as defined by meeting both of the following criteria: i. a "superscan" of bone scan, and ii. no soft tissue lesion that can be assessed by RECIST criteria
* Refractory nausea and vomiting, malabsorption syndrome, chronic gastrointestinal diseases, inability to swallow the formulated product or previous significant bowel resection, or other condition that would preclude adequate absorption of capivasertib
* Any other disease, metabolic dysfunction, physical examination finding, or clinical laboratory finding that, in the investigator's opinion, gives reasonable suspicion of a disease or condition that contra-indicates the use of an investigational drug, may affect the interpretation of the results, render the patient at high risk from treatment complications or interferes with obtaining informed consent
* Evidence of dementia, altered mental status, or any psychiatric condition that would prohibit understanding or rendering of informed consent
* Previous allogeneic bone marrow transplant or solid organ transplant
* History of another primary malignancy except for malignancy treated with curative intent with no known active disease ≥ 2 years before the first dose of study intervention and of low potential risk for recurrence. Exceptions include adequately resected non-melanoma skin cancer and curatively treated in situ disease.
* Treatment with any of the following:

  i. Nitrosourea or mitomycin C within 6 weeks of the first dose of study treatment ii. Any investigational agents or study drugs from a previous clinical study within 30 days or 5 half-lives (whichever is longer) of the first dose of study treatment iii. Any other chemotherapy, immunotherapy, immunosuppressant medication (other than corticosteroids) or anticancer agents within 3 weeks of the first dose of study treatment. A longer washout may be required for drugs with a long half-life (eg, biologics) iv. Strong inhibitors or strong inducers of CYP3A4 within 2 weeks before the start of study treatment (3 weeks for St John's wort). Note that adequate washout or dose reduction may be required for some CYP3A substrates prior to initiating Capivasertib dosing.
* Drugs known to significantly prolong the QT interval and associated with Torsades de Pointes within 5 half-lives of the first dose of study treatment
* Participation in another clinical study with an investigational product administered in the last 30 days or 5 half-lives, whichever is longer.
* History of hypersensitivity to active or inactive excipients of capivasertib, abiraterone, or drugs with a similar chemical structure or class.
* Involvement in the planning and/or conduct of the study (applies to both AstraZeneca staff and/or staff at the study site).
* Judgment by the investigator that the patient should not participate in the study if the patient is unlikely to comply with study procedures, restrictions and requirements.
* Any restriction or contraindication based on the local prescribing information that would prohibit the use of abiraterone.

Ages: 18 Years to 130 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1012 (Actual)
Dates: Start 2020-07-13 (Actual); Primary Completion 2024-10-07 (Actual); Study Completion 2027-03-29 (Estimated)

PRIMARY OUTCOMES:
Radiographic Progression-free Survival (rPFS) | Up to approximately 55 months
  rPFS is defined as the time from randomisation to radiographic progression, as assessed by the investigator per Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST) for soft tissue and/or Prostate Cancer Working Group 3 (PCWG3) for bone, or death due to any cause for each study arm.

SECONDARY OUTCOMES:
Overall survival (OS) | Up to approximately 80 months
  Overall survival is the length of time from randomisation until the date of death due to any cause.
Time to Start of First Subsequent Therapy or Death (TFST) | Up to approximately 55 months
  TFST is defined as time from randomisation to the earlier of: the start date of the first subsequent anticancer therapy after discontinuation of randomised treatment (capivasertib/placebo), or death due to any cause.
Symptomatic Skeletal Event-Free Survival (SSE-FS) | Up to approximately 80 months
  SSE-FS is defined as time from randomisation until any of the following: use of radiation therapy to prevent or relieve skeletal symptoms; Occurrence of new symptomatic pathological bone fractures (vertebral or non-vertebral); Occurrence of spinal cord compression; Orthopaedic surgical intervention for bone metastasis; Death due to any cause.
Time to Pain Progression (TTPP) | Up to approximately 80 months
  TTPP is defined as the time from randomisation to clinically meaningful pain progression base on a 2-point increase from baseline in the Brief Pain Inventory-Short Form (BPI-SF) Item 3 ("worst pain in 24 hours") score and/or initiation of/increase in opiate analgesic use.
Time to PSA progression | Up to approximately 55 months
  The time from randomisation to PSA progression, as determined by PCWG3 criteria.
Time To Castration Resistance (TTCR) | Up to approximately 80 months
  TTCR is defined as the time from randomisation to the first castration-resistant event (radiographic disease progression, PSA progression, or SSE), whichever occurs first, with castrate levels of testosterone (below 50 ng/dL).
Fatigue intensity, severity and interference domains assessed by the Brief Fatigue Inventory (BFI) | Up to approximately 80 months
  BFI endpoints may include: Time to deterioration in fatigue intensity; Time to deterioration in fatigue interference; Change from baseline in fatigue severity and fatigue interference domain scores.
Overall Pain Severity and Pain Interference as assessed by BPI-SF questionnaire | Up to approximately 80 months
  BPI-SF: Change from baseline in pain severity and pain interference domain scores.
Disease-Related Symptoms and HRQoL using the Functional Assessment of Cancer Therapy - Prostate Cancer (FACT-P) questionnaire | Up to approximately 80 months
  FACT-P endpoints may include: Time to deterioration in FACT-P scores; Change from baseline in FACT-P scores.
Progression-Free Survival after next-line treatment (PFS2) | Up to approximately 80 months
  PFS2 is defined as time from randomisation until progression on next-line treatment, as clinical progression, PSA progression, or radiographic progression determined by RECIST version 1.1 (soft tissue) and/or PCWG3 criteria (bone), as assessed by the investigator, or death due to any cause.
Plasma concentration of capivasertib pre-dose | Cycle 1 Day 15, Cycle 2 Day 1, Cycle 2 Day 15
Plasma concentration of capivasertib 1h post-dose | Cycle 1 Day 1
Plasma concentration of capivasertib 4h post-dose | Cycle 1 Day 1

OTHER OUTCOMES:
Incidence and Severity of Adverse Events (AEs) | Up to approximately 80 months
  Percentage of participants with an adverse event (AE), graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE), Version 5.0, including analysis of pre-specified AEs.
Systolic and diastolic blood pressure | Up to approximately 80 months
  millimetre or mercury (mmHg)
Pulse rate (heart rate) | Up to approximately 80 months
  Beats per minute (BPM)
Body Temperature | Up to approximately 80 months
  Celsius (°C)
Weight | Up to approximately 80 months
  Kilograms (kg)
Changes in Targeted Laboratory Results | Up to approximately 80 months
  Change from baseline in selected laboratory test results
QT interval (QTc) by electrical activity | Up to approximately 80 months
  Milliseconds (msec)

CONTACTS AND LOCATIONS:
Locations (263):
- United States (32):
  - Research Site, Tucson, Arizona
  - Research Site, La Jolla, California
  - Research Site, Orange, California
  - Research Site, San Diego, California
  - Research Site, Denver, Colorado
  - Research Site, Lakewood, Colorado
  - Research Site, Norwich, Connecticut
  - Research Site, Fort Myers, Florida
  - Research Site, West Palm Beach, Florida
  - Research Site, Chicago, Illinois
  - Research Site, Geneva, Illinois
  - Research Site, Lisle, Illinois
  - Research Site, Baltimore, Maryland
  - Research Site, Detroit, Michigan
  - Research Site, Grand Rapids, Michigan
  - Research Site, Troy, Michigan
  - Research Site, Syracuse, New York
  - Research Site, The Bronx, New York
  - Research Site, Asheville, North Carolina
  - Research Site, Durham, North Carolina
  - Research Site, Columbus, Ohio
  - Research Site, Lancaster, Pennsylvania
  - Research Site, Philadelphia, Pennsylvania
  - Research Site, Pittsburgh, Pennsylvania
  - Research Site, Charleston, South Carolina
  - Research Site, Myrtle Beach, South Carolina
  - Research Site, Chattanooga, Tennessee
  - Research Site, Houston, Texas
  - Research Site, Norfolk, Virginia
  - Research Site, Roanoke, Virginia
  - Research Site, Seattle, Washington
  - Research Site, Madison, Wisconsin
- Argentina (8):
  - Research Site, Berazategui
  - Research Site, Buenos Aires
  - Research Site, CABA
  - Research Site, Ciudad de Buenos Aires
  - Research Site, La Plata
  - Research Site, Mendoza
  - Research Site, Rosario
  - Research Site, San Salvador de Jujuy
- Australia (5):
  - Research Site, Birtinya
  - Research Site, Darlinghurst
  - Research Site, Kingswood
  - Research Site, Orange
  - Research Site, South Brisbane
- Austria (3):
  - Research Site, Graz
  - Research Site, Linz
  - Research Site, Salzburg
- Belgium (4):
  - Research Site, Anderlecht
  - Research Site, Ghent
  - Research Site, Kortrijk
  - Research Site, Liège
- Brazil (13):
  - Research Site, Belém
  - Research Site, Belo Horizonte
  - Research Site, Florianópolis
  - Research Site, Fortaleza
  - Research Site, Jaú
  - Research Site, Joinville
  - Research Site, Porto Alegre
  - Research Site, Ribeirão Preto
  - Research Site, Rio de Janeiro
  - Research Site, Santa Maria
  - Research Site, São José do Rio Preto
  - Research Site, São Paulo
  - Research Site, Três Lagoas
- Bulgaria (4):
  - Research Site, Pleven
  - Research Site, Plovdiv
  - Research Site, Sofia
  - Research Site, Varna
- Canada (8):
  - Research Site, Calgary, Alberta
  - Research Site, Edmonton, Alberta
  - Research Site, Kelowna, British Columbia
  - Research Site, Vancouver, British Columbia
  - Research Site, Brampton, Ontario
  - Research Site, Oshawa, Ontario
  - Research Site, Toronto, Ontario
  - Research Site, Montreal
- Chile (3):
  - Research Site, Santiago
  - Research Site, Temuco
  - Research Site, Viña del Mar
- China (22):
  - Research Site, Beijing
  - Research Site, Changchun
  - Research Site, Changsha
  - Research Site, Chengdu
  - Research Site, Chongqing
  - Research Site, Fuzhou
  - Research Site, Guangzhou
  - Research Site, Guiyang
  - Research Site, Hangzhou
  - Research Site, Kunming
  - Research Site, Nanchang
  - Research Site, Nanjing
  - Research Site, Nantong
  - Research Site, Ningbo
  - Research Site, Shanghai
  - Research Site, Shengyang
  - Research Site, Tianjin
  - Research Site, Wenzhou
  - Research Site, Wuhan
  - Research Site, Xi'an
  - Research Site, Yantai
  - Research Site, Zhengzhou
- Czechia (4):
  - Research Site, Brno
  - Research Site, Hořovice
  - Research Site, Hradec Králové
  - Research Site, Prague
- France (12):
  - Research Site, Besançon
  - Research Site, Bordeaux
  - Research Site, Marseille
  - Research Site, Montpellier
  - Research Site, Nice
  - Research Site, Paris
  - Research Site, Pierre-Bénite
  - Research Site, Quimper
  - Research Site, Rennes
  - Research Site, Strasbourg
  - Research Site, Suresnes
  - Research Site, Villejuif
- Germany (9):
  - Research Site, Berlin
  - Research Site, Duisburg
  - Research Site, Hamburg
  - Research Site, Herne
  - Research Site, Mettmann
  - Research Site, Münster
  - Research Site, Nuremberg
  - Research Site, Nürtingen
  - Research Site, Wesel
- Hong Kong (2):
  - Research Site, Hong Kong
  - Research Site, Lai Chi Kok
- India (14):
  - Research Site, Ahmedabad
  - Research Site, Bangalore
  - Research Site, Delhi
  - Research Site, Faridabad
  - Research Site, Kanpur
  - Research Site, Kolkata
  - Research Site, Madurai
  - Research Site, Manipal
  - Research Site, Meerut
  - Research Site, Mohali
  - Research Site, Nagpur
  - Research Site, New Delhi
  - Research Site, Thiruvananthapuram
  - Research Site, Varanasi
- Israel (6):
  - Research Site, Haifa
  - Research Site, Jerusalem
  - Research Site, Kfar Saba
  - Research Site, Petah Tikva
  - Research Site, Ramat Gan
  - Research Site, Ẕerifin
- Japan (34):
  - Research Site, Bunkyō City
  - Research Site, Chiba
  - Research Site, Chūōku
  - Research Site, Fukuoka
  - Research Site, Hamamatsu
  - Research Site, Hirakata-shi
  - Research Site, Hirosaki-shi
  - Research Site, Isehara-shi
  - Research Site, Kanazawa
  - Research Site, Kashihara-shi
  - Research Site, Kawagoe-shi
  - Research Site, Kisarazu-shi
  - Research Site, Kita-gun
  - Research Site, Kobe
  - Research Site, Kumamoto
  - Research Site, Kyoto
  - Research Site, Miyazaki
  - Research Site, Morioka
  - Research Site, Nagano
  - Research Site, Nagasaki
  - Research Site, Nagoya
  - Research Site, Natori-shi
  - Research Site, Osaka
  - Research Site, Osakasayama-shi
  - Research Site, Ota Shi
  - Research Site, Sagamihara-shi
  - Research Site, Sapporo
  - Research Site, Shinjuku-ku
  - Research Site, Toon-shi
  - Research Site, Tsu
  - Research Site, Ube-shi
  - Research Site, Yokohama
  - Research Site, Yokosuka-shi
  - Research Site, Yufu-shi
- Mexico (4):
  - Research Site, Culiacán
  - Research Site, Guadalajara
  - Research Site, Mexico City
  - Research Site, Monterrey
- Netherlands (6):
  - Research Site, Amsterdam
  - Research Site, Hilversum
  - Research Site, Roosendaal
  - Research Site, The Hague
  - Research Site, Tilburg
  - Research Site, Utrecht
- Peru (3):
  - Research Site, Callao
  - Research Site, Lima
  - Research Site, San Isidro
- Philippines (6):
  - Research Site, Baguio City
  - Research Site, Cebu City
  - Research Site, Davao City
  - Research Site, Iloilo City
  - Research Site, Quezon City
  - Research Site, San Juan City
- Poland (9):
  - Research Site, Bydgoszcz
  - Research Site, Gdansk
  - Research Site, Koszalin
  - Research Site, Lodz
  - Research Site, Olsztyn
  - Research Site, Poznan
  - Research Site, Rzeszów
  - Research Site, Torun
  - Research Site, Warsaw
- Russia (5):
  - Research Site, Moscow
  - Research Site, Novisibirsk
  - Research Site, Novosibirsk
  - Research Site, Saint Petersburg
  - Research Site, Yaroslavl
- Slovakia (6):
  - Research Site, Bratislava
  - Research Site, Martin
  - Research Site, Nitra
  - Research Site, Prešov
  - Research Site, Šaľa
  - Research Site, Trenčín
- South Africa (5):
  - Research Site, Cape Town
  - Research Site, Johannesburg
  - Research Site, Parow
  - Research Site, Port Elizabeth
  - Research Site, Pretoria
- South Korea (4):
  - Research Site, Daegu
  - Research Site, Goyang-si
  - Research Site, Seongnam-si
  - Research Site, Seoul
- Spain (7):
  - Research Site, Badalona (Barcelona)
  - Research Site, Barcelona
  - Research Site, Las Palmas de Gran Canaria
  - Research Site, Madrid
  - Research Site, Oviedo
  - Research Site, Santander
  - Research Site, Seville
- Taiwan (5):
  - Research Site, Kaohsiung City
  - Research Site, Taichung
  - Research Site, Tainan
  - Research Site, Taipei
  - Research Site, Taoyuan
- Thailand (5):
  - Research Site, Bangkok
  - Research Site, Chiang Mai
  - Research Site, Hat Yai
  - Research Site, Lampang
  - Research Site, Muang
- Turkey (Türkiye) (6):
  - Research Site, Ankara
  - Research Site, Antalya
  - Research Site, Eskişehir
  - Research Site, Istanbul
  - Research Site, Izmir
  - Research Site, Kayseri
- United Kingdom (6):
  - Research Site, Cambridge
  - Research Site, Guildford
  - Research Site, Manchester
  - Research Site, Plymouth
  - Research Site, Sutton
  - Research Site, Whitchurch
- Vietnam (3):
  - Research Site, Hanoi
  - Research Site, Hà Nội
  - Research Site, Ho Chi Minh City

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal Vivli.org. All request will be evaluated as per the AZ disclosure commitment:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure. "Yes", indicates that AZ are accepting requests for IPD, but this does not mean all requests will be approved.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA/PhRMA Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the de-identified individual patient-level data via secure research environment Vivli.org. A Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information.
URL: https://vivli.org/